CLINICAL TRIAL: NCT03383133
Title: Allosteric Regulation of Cytosolic Sulfotransferases in Humans
Brief Title: Studies of Sulfur Metabolism in Humans
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017-8685
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Metabolic Side Effects of Drugs
Keywords: sulfotransferase; metabolism; acetaminophen; dehydroepiandrosterone; mefenamic acid; allostery
MeSH Terms: conditions — Metabolic Side Effects of Drugs and Substances

STUDY DESIGN:
Intervention Model Description: This study will involve only a single individual.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SULT Allosteric Inhibition (Experimental): A single, therapeutic dose of acetaminophen (1.0 g)) or dehydroepiandrosterone (75 mg) is taken orally (with 375 ml of water) either alone or simultaneously with a single, oral, therapeutic dose of mefenamic acid (0.75 g).
  Interventions: Drug: SULT Allosteric Inhibition

INTERVENTIONS:
Drug: SULT Allosteric Inhibition — A single, therapeutic dose of acetaminophen (APAP, 1.0 g)) or dehydroepiandrosterone (DHEA, 75 mg) is taken orally (with 375 ml of water) either alone or simultaneously with a single, oral, therapeutic dose of mefenamic acid (MEF, 0.75 g). In total, 5 experiments will be performed. Each experiment is performed in duplicate. Compounds are taken prior to eating breakfast. One hour later, the patient has a light breakfast and eats normally thereafter. Urine samples are collected at 15', 30', 1 h, 2h, 3h, 4h, 5 h, 6h, 7h, 8h, 9h, 10h, 11h, and 12h intervals following dosing. The samples are weighed. A 10 ml aliquot is taken from each time point and the aliquots are stored at -20 °C. Samples (0.5 ml) are then transferred to NMR tubes spectra are taken to assess drug metabolites in urine.

SUMMARY:
The study test whether the NSAID allosteric site of human sulfotransferase 1A1 (SULT1A1) is operative in humans. The study will test the effects of mefenamic acid (MEF) on the sulfonation of acetaminophen (APAP, a SULT1A1 specific substrate) and dehydroepiandrosterone (DHEA, a SULT2A1 substrate). If the allosteric site is active in vivo, MEF is predicted to result in a decrease in sulfonation of APAP (MEF inhibits SULT with high affinity (Ki = 23 nM), and to have no effect on sulfonation of the DHEA (MEF has little or no effect on SULT2A1 activity).

DETAILED DESCRIPTION:
No patient registries associated with this study.

A single, therapeutic dose of acetaminophen (APAP, 1.0 g)) or dehydroepiandrosterone (DHEA, 75 mg) is taken orally (with 375 ml of water) either alone or simultaneously with a single, oral, therapeutic dose of mefenamic acid (MEF, 0.75 g). In total, 5 experiments will be performed: 1, APAP alone; 2, DHEA alone; 3, MEF alone; 4, APAP + MEF; and 5, DHEA + MEF. Each experiment will be performed in duplicate. Compounds will be taken prior to eating breakfast. One hour later, the patient has a light breakfast (Cheerios and milk, and a cup of coffee) and eats normally thereafter. Urine samples are collected at 15', 30', 1 h, 2h, 3h, 4h, 5 h, 6h, 7h, 8h, 9h, 10h, 11h, and 12h intervals following dosing. The study subject will attempt to completely empty their bladder at each urine-collection time point. The samples are weighed. A 10 ml aliquot is taken from each time point and the aliquots are stored at -20 °C. Samples (0.5 ml) are then transferred to nuclear magnetic resonance (NMR) tubes and NMR spectra are taken to assess drug metabolites in urine. Proton NMR will be performed using the 600 MHz instrument in the Einstein facility.

ELIGIBILITY:
Inclusion criteria:

* Gender - one male
* Age - 61 y.o.
* Healthy
* Agreed to sign the consent form

Exclusion criteria:

● None

Ages: 61 Years to 61 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Acetaminophen and Dehydroepiandrosterone Conjugates | 15min, 30min, 1hr, 2hr, 3hr, 4hr, 5hr, 6hr, 7hr, 8hr, 9hr, 10hr, 11hr, and 12hr following administration.
  Proton NMR Signals will be used to quantitate conjugates of acetaminophen and dehydroepiandrosterone in urine.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas S Leyh, Ph. D., Principal Investigator — The Albert Einstein College of Medicine
Locations (1):
- Albert Einstein Collage of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
This study will determine the levels acetaminophen and dehydroepiandrosterone conjugates in the urine of a single individuals. The levels will be published and

REFERENCES:
- [Background] Falany JL, Macrina N, Falany CN. Regulation of MCF-7 breast cancer cell growth by beta-estradiol sulfation. Breast Cancer Res Treat. 2002 Jul;74(2):167-76. doi: 10.1023/a:1016147004188. PMID 12186377
- [Background] Parker CR Jr. Dehydroepiandrosterone and dehydroepiandrosterone sulfate production in the human adrenal during development and aging. Steroids. 1999 Sep;64(9):640-7. doi: 10.1016/s0039-128x(99)00046-x. PMID 10503722
- [Background] Cook IT, Duniec-Dmuchowski Z, Kocarek TA, Runge-Morris M, Falany CN. 24-hydroxycholesterol sulfation by human cytosolic sulfotransferases: formation of monosulfates and disulfates, molecular modeling, sulfatase sensitivity, and inhibition of liver x receptor activation. Drug Metab Dispos. 2009 Oct;37(10):2069-78. doi: 10.1124/dmd.108.025759. Epub 2009 Jul 9. PMID 19589875
- [Background] Visser TJ. Role of sulfation in thyroid hormone metabolism. Chem Biol Interact. 1994 Jun;92(1-3):293-303. doi: 10.1016/0009-2797(94)90071-x. PMID 8033262
- [Background] Eisenhofer G, Coughtrie MW, Goldstein DS. Dopamine sulphate: an enigma resolved. Clin Exp Pharmacol Physiol Suppl. 1999 Apr;26:S41-53. PMID 10386253
- [Background] Swann J, Murry J, Young JA. Cytosolic sulfotransferase 1A1 regulates HIV-1 minus-strand DNA elongation in primary human monocyte-derived macrophages. Virol J. 2016 Feb 24;13:30. doi: 10.1186/s12985-016-0491-9. PMID 26906565
- [Background] Yalcin EB, More V, Neira KL, Lu ZJ, Cherrington NJ, Slitt AL, King RS. Downregulation of sulfotransferase expression and activity in diseased human livers. Drug Metab Dispos. 2013 Sep;41(9):1642-50. doi: 10.1124/dmd.113.050930. Epub 2013 Jun 17. PMID 23775849
- [Background] Wang T, Cook I, Leyh TS. The NSAID allosteric site of human cytosolic sulfotransferases. J Biol Chem. 2017 Dec 8;292(49):20305-20312. doi: 10.1074/jbc.M117.817387. Epub 2017 Oct 16. PMID 29038294
- [Background] Riches Z, Stanley EL, Bloomer JC, Coughtrie MW. Quantitative evaluation of the expression and activity of five major sulfotransferases (SULTs) in human tissues: the SULT "pie". Drug Metab Dispos. 2009 Nov;37(11):2255-61. doi: 10.1124/dmd.109.028399. Epub 2009 Aug 13. PMID 19679676
- [Background] Nagar S, Walther S, Blanchard RL. Sulfotransferase (SULT) 1A1 polymorphic variants *1, *2, and *3 are associated with altered enzymatic activity, cellular phenotype, and protein degradation. Mol Pharmacol. 2006 Jun;69(6):2084-92. doi: 10.1124/mol.105.019240. Epub 2006 Mar 3. PMID 16517757
- [Background] Falany CN, Vazquez ME, Kalb JM. Purification and characterization of human liver dehydroepiandrosterone sulphotransferase. Biochem J. 1989 Jun 15;260(3):641-6. doi: 10.1042/bj2600641. PMID 2764897
- [Background] Cook I, Wang T, Falany CN, Leyh TS. The allosteric binding sites of sulfotransferase 1A1. Drug Metab Dispos. 2015 Mar;43(3):418-23. doi: 10.1124/dmd.114.061887. Epub 2014 Dec 22. PMID 25534770
- [Background] Vietri M, De Santi C, Pietrabissa A, Mosca F, Pacifici GM. Inhibition of human liver phenol sulfotransferase by nonsteroidal anti-inflammatory drugs. Eur J Clin Pharmacol. 2000 Apr;56(1):81-7. doi: 10.1007/s002280050725. PMID 10853883